CLINICAL TRIAL: NCT02961777
Title: Study to Evaluate the Care Process and the Quality of Care for Adult Patients With ST Elevated Myocardial Infarction
Brief Title: Study to Evaluate the Care Process and the Quality of STEMI Care
Acronym: CP4ACS
Status: Completed | Type: Observational
Sponsor: European Pathway Association (Other)
Collaborators: KU Leuven (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Kris Vanhaecht, Professor, European Pathway Association
Other Study IDs: CP4ACS\2013\2
Record Dates: First submitted 2016-11-02; First posted 2016-11-11 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Myocardial Infarction; Acute Coronary Syndrome
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Time 1: retrospective evaluation of patient record. no intervention
- Time 2: retrospective evaluation of patient record. no intervention
  Interventions: Other: implementation of care pathway
- Time 3: retrospective evaluation of patient record. no intervention
  Interventions: Other: implementation of care pathway

INTERVENTIONS:
Other: implementation of care pathway — implementation of a care pathway
  Groups: Time 2; Time 3

SUMMARY:
Cardiovascular diseases, and more precisely patients with ST - elevated myocardial infarction are globally responsible for a large number of hospitalizations and deaths. Monitoring the quality of care for these patients is very relevant topic. Investigators developed indicators from the scientific literature on the quality of care for patients with STEMI at both the patient level and hospital level. The indicators were subsequently validated by a RAND modified Delphi - study of multidisciplinary experts in the care of patients with STEMI.

In this study, the following objectives are set:

1. ) Study of the quality of care for patients with STEMI in 16 Flemish hospitals with cardiology department by retrospective and prospective audit of 20 patient records per participating hospital .
2. ) Study of the interdisciplinary relationships and communication within teams involved in the care of patients with STEMI in the participating hospitals 3) Study of perceived organization of care for patients with STEMI in the participating hospitals

In accordance with the objectives of the research, the study consists of three phases:

1. ) A retrospective observational audit of 20 patient records of patients with STEMI each participating hospital.
2. ) A prospective observational audit of 20 patient records of patients with STEMI each participating hospital.
3. ) A survey using validated instruments of interdisciplinary relationships and communication on the one hand and on the other by the teams involved in the care of patients with STEMI perceived organization of care .

Data collection is performed by local researchers and remains their property. The data is coded and kept confidential. Only the local researcher has access to the encryption key. The data are protected by the Belgian law on privacy and medical confidentiality, only to be used in the context of this study. The results are published anonymously.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted with STEMI within 24 hours after symptom onset and
* eligible for reperfusion according to ESC STEMI guidelines

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted with STEMI within 24 hours after symptom onset and eligble for reperfusion according to ESC STEMI guidelines
Sampling Method: Probability Sample
Enrollment: 640 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
performance on quality indicators at patient level as defined by the CP4ACS Delphi Study to Determine Appropriateness of STEMI Quality Indicators in Belgium (NCT02030210) | through study completion, an average of 1 year
  This study evaluates quality indicators at patient level as defined by the CP4ACS Delphi Study to Determine Appropriateness of STEMI Quality Indicators in Belgium. The study is limited to the period in which the patients are hospitalized; No data is gathered before or after hospitalization.
performance on quality indicators at hospital level as defined by the CP4ACS Delphi Study to Determine Appropriateness of STEMI Quality Indicators in Belgium (NCT02030210) | through study completion, an average of 1 year
  This study evaluates quality indicators at hospital level as defined by the CP4ACS Delphi Study to Determine Appropriateness of STEMI Quality Indicators in Belgium. The study is limited to the period in which the patients are hospitalized. No data is gathered before or after hospitalization.

IPD SHARING:
Plan to Share IPD: No